CLINICAL TRIAL: NCT03555409
Title: Clinical Feature and Treatment of Microsporidial Keratoconjunctivitis
Acronym: MKC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805063RINA
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Microsporidial Keratoconjunctivitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project was to analysis the causes, pathogenesis, diagnostic modalities and treatment outcomes of microsporidial keratoconjunctivitis.

DETAILED DESCRIPTION:
Microsporidia comprise a diverse group of obligate spore-forming intracellular eukaryotic pathogens first described in immunocompromised patients. Many species of microsporidia are found in aquatic environments, and they are considered as waterborne pathogens.Microsporidia are opportunistic pathogens that are reported to cause infections in various organs, including the eyes. The ocular appearance of this infection can manifest as corneal stromal keratitis or a superficial punctate keratoconjunctivitis. In particular, the characteristic feature of microsporidial keratoconjunctivitis is multiple whitish, slightly elevated epithelial lesions in conjunction with acute conjunctivitis. Awareness of microsporidial keratoconjunctivitis is increasing, and the number of cases reported is on the rise. This study was a retrospective case series of patients diagnosed as microsporidial keratoconjunctivitis. The purpose of this project was to analysis the causes, pathogenesis, diagnostic modalities and treatment outcomes of microsporidial keratoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as microsporidial keratoconjunctivitis

Exclusion Criteria:

* Patients diagnosed as bacterial or viral keratoconjunctivitis

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Microsporidia keratoconjunctivitis diagnosed at the National Taiwan University Hospital (NTUH)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Full chart records of the patients who diagnosed as microsporidial keratoconjunctivitis | 2018/6/1-2019/5/31
  Charts of all patients diagnosed as microsporidial keratoconjunctivitis between January, 2008 and April, 2018 at National Taiwan University Hospital were reviewed.

CONTACTS AND LOCATIONS:
Overall Officials: I-Jong Wang, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan